CLINICAL TRIAL: NCT00892216
Title: Does Acupressure Decrease Post-operative Nausea and Vomiting After the NUSS Procedure?
Brief Title: Does Acupressure Decrease Post-operative Nausea and Vomiting (PONV) After the Pectus Excavatum Correction (NUSS) Procedure?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants for study to be completed
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-188
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Pectus Excavatum
Keywords: PONV; NUSS procedure; Acupressure; Pectus Excavatum
MeSH Terms: conditions — Funnel Chest; Postoperative Nausea and Vomiting | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupressure Band (Experimental): A band with bead attachment will be used to produce Acupressure and applied to the P6 (three fingers breath from the wrist crease on th ventral surface of the upper limb). The application will be done 20 minutes prior to anesthesia and explanation as to usage after surgery will be given. The patient of caregiver will apply pressure on the bead for three minutes and repeat this four times a day for the next five days. None of the protocol for prevention of PONV in this group of patients will be changed. The postoperative therapy for nausea and vomiting will be on a PRN (as required) basis. Nausea and vomiting scores and VAS scores for pain estimation will be carried out according to hospital protocol in the PACU amd twice a day thereafter for their period of stay in the hospital. The amount of analgesics and antiemetics used and the number of days spent in the hospital will be registered.
  Interventions: Device: Acupressure (BioBand)
- Sham Acupressure (Sham Comparator): The same band will be placed and turned so the beads face the corresponding point on the dorsal surface of the upper limb area.
  Interventions: Device: Acupressure (BioBand)

INTERVENTIONS:
Device: Acupressure (BioBand) — Band will remain on from 20 minutes before surgery until the end of the hospital stay.
  Other Names: BioBand
  Arms: Acupressure Band
Device: Acupressure (BioBand) — Band will remain on from 20 minutes before surgery until the end of the hospital stay. The same band will be placed and turned so the beads face the corresponding point on the dorsal surface of the upper limb area.
  Other Names: BioBand
  Arms: Sham Acupressure

SUMMARY:
Post-operative nausea and vomiting (PONV) is not only unpleasant for patients but also can delay hospital discharge and increase cost of stay. In some cases, when severe vomiting occurs, pain scores seem to be increased. The overall incidence of PONV is 30% and increases to 79% in patients at high risk for this post-operative outcome. The NUSS procedure is considered to be a procedure with a high risk for the outcome of nausea and vomiting.

DETAILED DESCRIPTION:
The rationale is to do a prospective study in patients who have been diagnosed with Pectus Excavatum and who are undergoing a NUSS procedure (pectus excavatum correction) and to evaluate the effect of Acupressure on the post-operative outcome of PONV in these patients. Also, to determine whether there are any secondary outcomes related to pain scores and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* age 8-40 years old
* ASA 1-3
* males & females

Exclusion Criteria:

* local infection of the site - P6
* acupuncture treatment within 8 weeks of the preoperative period
* coagulopathy is a contraindication for Acupuncture but not Acupressure

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2005-04; Primary Completion 2010-01 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Relief of PONV. This effect will be evaluated in the PACU and then twice a day until discharge which is usually 5 days post-operative. Hospital score for nausea and vomiting will be used. | Twice a day for 5 days

SECONDARY OUTCOMES:
Possibility of decrease in VAS score and hospital stay when compared to control group. | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Meena Nandagopal, M.B.B.S. DLO, DARCS, FFARCS(I), Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- McMaster University Hospital, HHSC/Hamilton Health Sciences, Hamilton, Ontario, Canada